CLINICAL TRIAL: NCT01525524
Title: Treatment of Major Depressive Disorder Post Stroke With Transcranial Direct Current Stimulation (TDCS): Randomized, Double-Blind, Clinical Trial
Brief Title: Treatment of Major Depressive Disorder Post Stroke With Transcranial Direct Current Stimulation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Leandro Valiengo, Principal Investigator, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1180/12
Record Dates: First submitted 2012-01-24; First posted 2012-02-03 (Estimated); Last update posted 2014-09-09 (Estimated); Status verified 2014-09

CONDITIONS: Major Depressive Disorder 1
Keywords: tDCS; Major Depression; Stroke
MeSH Terms: conditions — Major Depressive Disorder 1; Depressive Disorder, Major; Stroke | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sham Stimulation (Sham Comparator): In active stimulation, the anode is placed over the left dorsolateral prefrontal cortex and the cathode is placed over the right prefrontal cortex with the Transcranial Direct Current Stimulation. They are located five centimeters ventrally of the primary motor area, which are located five centimeters laterally of the central point of the scalp. The device will deliver a charge of 2mA for 1 minute, after that the device will be automatically turned off for 29 minutes.
  Interventions: Device: Transcranial Direct Current Stimulation
- Active Stimulation (Active Comparator): In active stimulation, the anode is placed over the left dorsolateral prefrontal cortex and the cathode is placed over the right prefrontal cortex with the transcranial Direct Current Stimulation device. They are located five centimeters ventrally of the primary motor area, which are located five centimeters laterally of the central point of the scalp. The device will deliver a charge of 2mA for 30 minutes.
  Interventions: Device: Transcranial Direct Current Stimulation

INTERVENTIONS:
Device: Transcranial Direct Current Stimulation — In active stimulation(active Transcranial Direct Current Stimulation), the anode is placed over the left dorsolateral prefrontal cortex and the cathode is placed over the right prefrontal cortex. They are located five centimeters ventrally of the primary motor area, which are located five centimeters laterally of the central point of the scalp (which is located on the intersection of the sagittal and median curves). The device will deliver a charge of 2mA for 30 minutes.
  Other Names: Transcranial Stimulation

SUMMARY:
Stroke is one of the main public health problems in America Latina. It can be associated with several neuropsychiatric complications, which include a broad spectrum of emotional distress and cognitive, results in important clinical implications for the prognosis of these patients. Depression is a common complication, affecting around 5-72% of patients and is associated with various cognitive deficits and also with increased mortality - up to 50% more deaths compared to non-depressed patients. Treatment of depression after stroke is important not only to improve depressive symptoms but can also be beneficial for cognitive deficits, activities of daily living. and leads to increased survival for these patients. There are different treatments for depression after stroke, all showing inconclusive results, even though antidepressants have been effective in some groups of patients, tolerability and treatment adherence were not very good-so it is necessary that new therapeutic modalities are presented with good tolerability. In this sense, transcranial direct current stimulation (tDCS) is an interesting technique that can provide interesting results, which proved to be effective for depression in some studies. This study proposes to investigate the effect of tDCS for the treatment of major depressive disorder after stroke. The proposed design is a clinical trial, randomized, double-blind, placebo-controlled study in a subsample of participants in the prospective cohort of stroke: Study of Morbidity and Mortality of stroke. They will be allocated to one of the groups: sham or active tDCS group. Participants will receive ten consecutive days of active or sham stimulation and return at the end of two weeks to evaluate the improvement in depression, cognition and functionality. As objectives, the investigators expect to see a clinical improvement of depression through scales like Hamilton, Beck and MADRS(Montgomery-Asberg Depression Rating Scale), and expect improvement on cognitive tests as MoCA (Montreal Cognitive Assessment), MMSE (mini mental scale exam), FAB (frontal assessment battery) and trail test. Another goal is to see improvement in markers related to depression as BDNF, cortisol, interleukins and heart rate variability. With all this, the investigators hope to offer a new treatment, and effective with few side effects to treat depression after stroke.

DETAILED DESCRIPTION:
The Study of Morbidity and Mortality of stroke (EMMA) is a cohort study of patients with stroke.

ELIGIBILITY:
Inclusion Criteria:

* Major Depressive Disorder after stroke
* First episode of Stroke
* Hamilton > 17

Exclusion Criteria:

* Others severe neurologic conditions
* Others Axis I besides anxiety
* Important suicidal ideation
* Use of antidepressants

Ages: 30 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2012-01; Primary Completion 2013-12 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Treatment response | Week 4 after tenth day of tDCS
  Hamilton of active will be lower than sham group

SECONDARY OUTCOMES:
Treatment response | Week 4 after tenth day of tDCS
  Response is defined as less than 50% of baseline Hamilton

CONTACTS AND LOCATIONS:
Overall Officials: Leandro Valiengo, MD, Principal Investigator — HU-USP
Locations (1):
- University of Sao Paulo, São Paulo, São Paulo, Brazil

REFERENCES:
- [Derived] Valiengo LC, Goulart AC, de Oliveira JF, Bensenor IM, Lotufo PA, Brunoni AR. Transcranial direct current stimulation for the treatment of post-stroke depression: results from a randomised, sham-controlled, double-blinded trial. J Neurol Neurosurg Psychiatry. 2017 Feb;88(2):170-175. doi: 10.1136/jnnp-2016-314075. Epub 2016 Nov 4. PMID 27815324